CLINICAL TRIAL: NCT01064505
Title: A Phase I Open-Label, Dose Escalation Trial of QPI-1007 Delivered by a Single Intravitreal Injection to Patients With Optic Nerve Atrophy (Stratum I) and Acute Non-Arteritic Anterior Ischemic Optic Neuropathy (NAION) (Stratum II)
Brief Title: Safety Study of a Single IVT Injection of QPI-1007 in Chronic Optic Nerve Atrophy and Recent Onset NAION Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Quark Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: QRK.007
Record Dates: First submitted 2010-02-04; First posted 2010-02-08 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2013-05

CONDITIONS: Optic Atrophy; Non-arteritic Anterior Ischemic Optic Neuropathy
Keywords: Ocular Neuroprotection; ocular neuroprotectant; NAION; NAAION; Non-arteritic ischemic optic neuropathy; Non-arteritic anterior ischemic optic neuropathy; chronic optic nerve atrophy; optic nerve atrophy; retinal degeneration; optic neuritis; end stage glaucoma; Leber's hereditary optic neuropathy
MeSH Terms: conditions — Optic Atrophy; Optic Neuropathy, Ischemic; Retinal Degeneration; Optic Neuritis; Optic Atrophy, Hereditary, Leber | interventions — RNA, Small Interfering

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- QPI-1007 (Experimental)
  Interventions: Drug: QPI-1007 at various doses

INTERVENTIONS:
Drug: QPI-1007 at various doses — Single Intravitreal Injection
  Other Names: QPI-1007; siRNA; small interfering RNA; short interfering RNA

SUMMARY:
This is an open-label, dose escalation, safety, tolerability and pharmacokinetic study, where active study drug (QPI-1007) will be given to all patients who participate.

This study will determine whether QPI-1007 is safe when it is injected into the eye. The study will also reveal if there are any side effects of the drug and how long it takes for the body to clear the drug.

DETAILED DESCRIPTION:
Patients will be enrolled according to one of two sets of criteria designated as Stratum I and Stratum II.

1. Stratum I will enroll Optic Nerve Atrophy patients who meet necessary criteria. Stratum I will consist of a maximum of 6 cohorts and each cohort will enroll 3 to 6 evaluable patients. Enrollment in Stratum I is now closed.
2. Stratum II will enroll patients diagnosed with acute Non Arteritic Anterior Ischemic Optic Neuropathy (NAION) within 28 days of symptom onset who meet necessary criteria. Stratum II will consist of a maximum of 3 cohorts and each cohort will enroll up to 10 evaluable patients. Enrollment in Stratum II is still open.

ELIGIBILITY:
Key Stratum I (Chronic Optic Nerve Atrophy) Inclusion Criteria:

* "Legally blind" in the study eye as the result of an irreversible condition affecting the posterior segment of the eye.
* Clear ocular media and able to undergo adequate pupil dilation.
* Visual acuity and visual field in the non-study eye are better than or equal to the study eye
* At least 21 years old.

Key Stratum I (Chronic Optic Nerve Atrophy) Exclusion Criteria:

* For the study eye only: history of any IVT injection or vitrectomy, vitreous hemorrhage, retinal detachment, or active inflammatory condition (e.g. conjunctivitis).
* For either eye: history of uveitis.

Enrollment is now closed in Stratum I.

Key Stratum II (Acute NAION) Inclusion Criteria:

* Positive diagnosis of NAION with symptom onset within 28 days prior to planned dosing with QPI-1007.
* Visual acuity in the study eye is between 20/40 and light perception.
* Clear ocular media and able to undergo adequate pupil dilation.
* At least 50 years old.

Key Stratum II (Acute NAION) Exclusion Criteria:

* For the study eye only: Macular disease, retinopathy, or other eye disease limiting visual acuity; prior intraocular surgery (other than Lasik) and cataract surgery within 3 months prior to dosing; glaucoma laser surgery within 1 month prior to dosing; pain on or aggravated by eye movement; history of vitreous hemorrhage; history of retinal detachment; any active inflammatory condition (e.g. conjunctivitis); glaucoma or ocular hypertension; or intraocular pressure > 26 mmHg.
* For either eye: History of optic neuritis; or history of uveitis.
* Received any treatment for NAION prior to dosing.
* Any other abnormality which in the opinion of the investigator is suggestive of a disease other than NAION in the study eye only.
* Clinical evidence of temporal arteritis.
* History of collagen vascular disease or other inflammatory disease, or history of multiple sclerosis.

Enrollment in Stratum II is still open.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2010-02; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
To determine the safety, tolerability and the dose-limiting toxicities (DLTs) of QPI 1007 when administered as a single intravitreal (IVT) injection. | 12 Months Post-injection
To assess the pharmacokinetics (PK) of QPI-1007 when administered as a single IVT injection. | 12 Months Post-Injection

SECONDARY OUTCOMES:
To determine the presence of and to describe any anatomical changes in the optic nerve head and retina observed following the administration of a single IVT injection of QPI 1007. | 12 Months Post-Injection
To assess any changes in visual acuity and visual field observed following the administration of a single IVT injection of QPI-1007. | 12 Months Post-Injection

CONTACTS AND LOCATIONS:
Overall Officials: Rabia Ozden, MD, Study Director — Quark Pharmaceuticals
Locations (28):
- United States (22):
  - Retinal Consultants of Arizona, Phoenix, Arizona
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - Jules Stein Eye Institute, University of California, Los Angeles, Los Angeles, California
  - Rocky Mountain Multiple Sclerosis Center at Anschutz Medical Campus, University of Colorado, Aurora, Colorado
  - Bascom Palmer at the University of Miami, Miami, Florida
  - Sarasota Retina Institute, Sarasota, Florida
  - University of Illinois at Chicago, Eye and Ear Infirmary, Chicago, Illinois
  - Kansas University Medical Center, Kansas City, Kansas
  - University of Kentucky, Department of Ophthalmology, Lexington, Kentucky
  - University of Minnesota, Department of Ophthalmology, Minneapolis, Minnesota
  - Mason Eye Institute, University of Missouri, Columbia, Missouri
  - New York Eye and Ear Infirmary, New York, New York
  - Flaum Eye Institute, University of Rochester Medical Center, Rochester, New York
  - Western Carolina Retinal Associates, Asheville, North Carolina
  - Charlotte Eye, Ear, Nose and Throat Associates, PA, Charlotte, North Carolina
  - Duke Eye Center, Duke University Medical Center, Durham, North Carolina
  - Cole Eye Institute, Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pennsylvania, Department of Ophthalmology, Philadelphia, Pennsylvania
  - Allegheny Ophthalmic and Orbital Associates, Pittsburgh, Pennsylvania
  - Alkek Eye Center Baylor College of Medicine, Houston, Texas
  - John A. Moran Eye Center at the University of Utah, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
- Israel (6):
  - Soroka University Medical Center, Dept of Ophthalmology, Beersheba
  - Bnai Zion Medical Center, Haifa
  - Rabin Medical Center, Belinson Campus, Dept of Ophthalmology, Petah Tikva
  - Kaplan Medical Center, Department of Ophthalmology, Rehovot
  - The Tel-Aviv Sourasky Medical Center, Dept of Ophthalmology, Tel Aviv
  - The Chaim Sheba Medical Center, Dept of Ophthalmology, Tel Litwinsky